CLINICAL TRIAL: NCT02864758
Title: Benefit-Risk Of Arterial THrombotic prEvention With Rivaroxaban for Atrial Fibrillation in Daily Clinical Practice - A French Cohort Within the Nationwide Claims and Hospital Database
Brief Title: Benefit-Risk Of Arterial THrombotic prEvention With Rivaroxaban for Atrial Fibrillation in France
Acronym: BROTHER
Status: Completed | Type: Observational
Sponsor: Bayer (Industry)
Collaborators: Janssen Scientific Affairs, LLC (Industry)
Responsible Party: Sponsor
Other Study IDs: 18656
Record Dates: First submitted 2016-08-09; First posted 2016-08-12 (Estimated); Last update posted 2023-11-07 (Actual); Status verified 2023-11

CONDITIONS: Atrial Fibrillation
MeSH Terms: conditions — Atrial Fibrillation | interventions — Rivaroxaban; acarboxyprothrombin; Dabigatran

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Group 1: Adult patients with nonvalvular atrial fibrillation (NVAF) treated with rivaroxaban
  Interventions: Drug: Rivaroxaban (Xarelto, BAY59-7939)
- Group 2: Adult patients with nonvalvular atrial fibrillation (NVAF) treated with vitamin k anatognists
  Interventions: Drug: Vitamin K antagonists
- Group 3: Adult patients with nonvalvular atrial fibrillation (NVAF) treated with dabigatran
  Interventions: Drug: dabigatran (Pradaxa)

INTERVENTIONS:
Drug: Rivaroxaban (Xarelto, BAY59-7939) — Tablets, 20mg once daily
  Groups: Group 1
Drug: Vitamin K antagonists — Tablets, dose is based on International Normalized Ratio
  Groups: Group 2
Drug: dabigatran (Pradaxa) — Tablets, 150 mg twice daily
  Groups: Group 3

SUMMARY:
The purpose of the study is to compare the one-year and two-year risk of each of the following individual outcomes: Stroke and systemic embolism (SE), major bleeding and death between new users of anticoagulant for Stroke prevention in atrial fibrillation (SPAF) during drug exposure: rivaroxaban versus Vitamin K antagonists (VKA), and rivaroxaban versus dabigatran

DETAILED DESCRIPTION:
Main objective: To compare the one-year and two-year risk of each of the following individual outcomes: Stroke and systemic embolism (SE), major bleeding and death between new users of anticoagulant for SPAF during drug exposure: rivaroxaban versus VKA, and rivaroxaban versus dabigatran.

Secondary objectives:

* To describe the drug exposure to rivaroxaban, dabigatran, and VKA for SPAF in new users, as well as and pattern of use;
* To compare the one-year and two-year risk of the following individual outcomes: a composite of stroke and SE, major bleeding and death, clinically relevant bleeding (CRB) and acute coronary syndrome (ACS) between new users of anticoagulant for SPAF during drug exposure: rivaroxaban versus VKA, and rivaroxaban versus dabigatran;
* To estimate the cumulative incidence and the incidence rate of each individual main and secondary outcome (stroke and SE, major bleeding, CRB, death, composite criteria, and ACS), as well as according to individual diagnose of each of these outcomes, during drug exposure for rivaroxaban, dabigatran, and VKA;
* To estimate the cumulative incidence of each individual main and secondary outcome (stroke and SE, major bleeding, CRB, death, composite criteria, and ACS), as well as according individual diagnose of each of these outcomes during post-anticoagulant exposure for rivaroxaban, dabigatran, and VKA (i.e. after anticoagulant discontinuation);
* To assess outcome risk factors, including (but not limited to), gender, age, stroke and bleeding risk scores (CHA2DS2-VASc and HAS-BLED), low or high dosage at index date for DOAC, drug predisposing to bleeding during drug exposure and significant baseline characteristics;
* To describe and compare healthcare resources utilisation related to SPAF during rivaroxaban, dabigatran, and VKA exposure, including outcomes, and their related costs from the societal perspective and from the French healthcare insurance perspective.

ELIGIBILITY:
Inclusion Criteria:

* Definite non-valvular atrial fibrillation:
* A first reimbursed dispensation of rivaroxaban, dabigatran, or VKA in 2013 or 2014, and
* No previous DOAC (rivaroxaban, dabigatran, apixaban) or VKA dispensation during the previous three years,
* Definite AF information in the database Probable non-valvular atrial fibrillation:-
* A first reimbursed dispensation of rivaroxaban, dabigatran, or VKA in 2013 or 2014, and
* No previous DOAC (rivaroxaban, dabigatran, apixaban) or VKA dispensation during the previous three years,
* Probable AF information in the database (using the development of an AF disease score, see variables definition below),

Exclusion Criteria:

* Patients with Rheumatic valve disease
* Patients with valve replacement
* Patients treated with anticoagulants for venous
* thromboemboslim or prevention of venous
* thromboembolism after orthopedic surgery

Ages: 2 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All subjects with a first reimbursed dispensation of rivaroxaban (15 or 20 mg), dabigatran (110 or 150 mg) or vitamin k antagonists in 2013 or 2014 diagnosed with Atrial Fibrillation
Sampling Method: Non-Probability Sample
Enrollment: 99999 (Actual)
Dates: Start 2016-09-08 (Actual); Primary Completion 2018-09-30 (Actual); Study Completion 2018-09-30 (Actual)

PRIMARY OUTCOMES:
Stroke and systemic embolism (Effectiveness outcome) | One year and Two Year
  Hospitalization with ischemic or undefined stroke or other systemic arterial embolism or surgical procedure for systemic arterial embolism To compare one year and two year risk between new users of anticoagulant for SPAF during drug exposure: rivaroxaban versus VKA, and rivaroxaban versus dabigatran.
Major Bleeding | One year and Two Year
  Hospitalization with haemorrhagic stroke, other critical organ or site bleeding (intraspinal, intraocular,retroperitoneal, intraarticular or pericardial, or intramuscular), Other bleeding with a transfusion during hospital stay, or resulting in death.
  To compare one year and two year risk between new users of anticoagulant for SPAF during drug exposure: rivaroxaban versus VKA, and rivaroxaban versus dabigatran.
Death | One year and Two Year
  All-cause death. To compare one year and two year risk between new users of anticoagulant for SPAF during drug exposure: rivaroxaban versus VKA, and rivaroxaban versus dabigatran.

SECONDARY OUTCOMES:
Pattern of use (Exposure, Adherence, Discontinuation, Switch) | Up to two years
  To describe the drug exposure to rivaroxaban, dabigatran, and VKA for SPAF in new users and pattern of use
A composite of stroke and SE, major bleeding and death, clinically relevant bleeding and acute coronary syndrome | One year and Two Year
  To compare one year and two year risk between new users of anticoagulant for SPAF during drug exposure: rivaroxaban vs VKA, and rivaroxaban vs dabigatran
Cumulative incidence and incidence rate of stroke and SE, major bleeding, clinically relevant bleeding, death, composite criteria, and acute coronary syndrome as well as according individual diagnose of each of these outcomes | Up to two years
  During drug exposure for rivaroxaban, dabigatran, and VKA
Cumulative incidence of Stroke and SE, major bleeding, clinically relevant bleeding, death, composite criteria, and acute coronary syndrome as well as according individual diagnose of each of these outcomes | Up to two years
  Post-anticoagulant exposure for rivaroxaban, dabigatran, and VKA (i.e. after anticoagulant discontinuation)
Healthcare resources utilisation | Up to two years
  Healthcare resources use will be described from reimbursed claims and hospitalisation information Healthcare resources cost will be estimated using the French HAS methodological guide for economic evaluations (2011)

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (1):
- Many Locations, Multiple Locations, France

REFERENCES:
- [Background] Blin P, Fauchier L, Dureau-Pournin C, Sacher F, Dallongeville J, Bernard MA, Lassalle R, Droz-Perroteau C, Moore N. Effectiveness and Safety of Rivaroxaban 15 or 20 mg Versus Vitamin K Antagonists in Nonvalvular Atrial Fibrillation. Stroke. 2019 Sep;50(9):2469-2476. doi: 10.1161/STROKEAHA.119.025824. Epub 2019 Aug 8. PMID 31390972
- [Derived] Fauchier L, Blin P, Sacher F, Dureau-Pournin C, Bernard MA, Lassalle R, Droz-Perroteau C, Dallongeville J, Moore N. Reduced dose of rivaroxaban and dabigatran vs. vitamin K antagonists in very elderly patients with atrial fibrillation in a nationwide cohort study. Europace. 2020 Feb 1;22(2):205-215. doi: 10.1093/europace/euz285. PMID 31638652